CLINICAL TRIAL: NCT01134627
Title: A Multi-centre, Double Blind, Randomized, Placebo Controlled, Parallel Group Trial Investigating Minocycline Versus Placebo as Add-on Therapy in Patients Who Are on Treatment With Interferon-beta-1a 44 Mcg Tiw (Rebif®) for the Treatment of Relapsing-Remitting Multiple Sclerosis
Brief Title: Minocycline as add-on to Interferon Beta-1a [IFN Beta-1a] (Rebif®) in Relapsing-Remitting Multiple Sclerosis [RRMS]
Acronym: RECYCLINE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMP 26588; 2005-004289-18 (EudraCT Number); NCT00381459 (obsolete NCT alias)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Interferon-β; Rebif®; Minocycline
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline group (Experimental)
  Interventions: Drug: Minocycline
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline — Participants who are self-administering Rebif® (IFN beta-1a) 44 microgram (mcg) as subcutaneous (sc) injection thrice weekly will also receive minocycline 100 milligram (mg) tablet twice daily as an add-on therapy in accordance with clinical practice for 96 weeks.
  Arms: Minocycline group
Drug: Placebo — Participants who are self-administering Rebif® (IFN beta-1a) 44 mcg as sc injection thrice weekly will also receive placebo tablets twice daily for 96 weeks.
  Arms: Placebo Group

SUMMARY:
This is a multicentric, double-blind, placebo-controlled, randomized, parallel group study to estimate the effect of minocycline as add-on to interferon beta-1a (IFN beta-1a) in subjects with relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
Interferon beta-1a is the approved standard therapy in RRMS. The beneficial effects of minocycline in the experimental autoimmune encephalomyelitis (EAE) model and its possible inhibitory effect on the degradation of IFN beta-1a suggest that minocycline treatment may have beneficial effects in MS as add-on therapy in subjects who are on treatment with IFN beta-1a. Adjuvant treatment with minocycline is easy to administer, well tolerated and relatively inexpensive. This is a multicentric, double blind, placebo controlled, randomized, parallel group study. Eligible subjects already started with IFN beta-1a (Rebif®) will be randomized 1:1 for treatment with either minocycline 2*100 mg daily as add-on therapy or placebo. The subjects will be examined clinically at baseline and after 12, 24, 48, 72 and 96 weeks. Laboratory tests (hematology and clinical chemistry) will be performed at baseline and after 4, 8, 12, 24, 36, 48, 60, 72, 84 and 96 weeks (at 4, 8, 36, 60 and 84 weeks only an additional liver enzyme test will be scheduled). The MRI (T1-weighted and T2-weighted) before treatment and after 96 weeks and immunological studies before treatment and after 48 weeks will be performed in a limited number of subjects in selected centers.

OBJECTIVES

Primary Objective:

The effect of minocycline versus placebo in subjects receiving treatment with IFN beta-1a on the time to the first documented relapse

Secondary Objectives:

* To estimate the effect of minocycline versus placebo in subjects receiving treatment with IFN beta-1a on the mean number of documented relapses per subject up to year 2
* To estimate, in a limited number of 120 subjects at pre-selected sites, the effect of minocycline versus placebo in subjects receiving treatment with IFN beta-1a on the number of new or enlarging lesions on T2-weighted MRI, changes in brain volume measured on MRI

Tertiary Objectives:

* Time to onset of disability progression sustained over at least 6 months based on change from baseline in EDSS in subjects with RRMS who recently started treatment with IFN beta-1a. (Disability progression is defined as an increase of: 1.0 point on the EDSS if EDSS was >= 1.0 at baseline; and 1.5 point on the EDSS if EDSS was 0.0 at baseline)
* Time to sustained progression by 2 points in 1 Functional System or 1 point in 2 Functional Systems
* The total number of reported relapses (documented and undocumented). An undocumented relapse is defined as the appearance of new symptoms or worsening of an old symptom, in the absence of fever, over at least 24 hours that could be attributed to MS activity, preceded by stability or improvement for at least 30 days
* The requirement for treatment with glucocorticoids due to relapses
* The time to first relapse
* The number of relapse-free (documented and undocumented relapses) subjects without progression
* The disease activity measured on the integrated disability status scale (IDSS)
* The number of subjects with a permanent loss of disability of 1.0 score on the EDSS, confirmed at 2 consecutive visits with an interval of 6 months
* The total area of MS lesions on T1 and T2-weighted MRI
* Analyze the safety with respect to the combination of Rebif® and minocycline
* Rate of dose reduction of IFN beta-1a (Rebif®)
* Relapse severity based on the EDSS and IDSS
* Immunological analyses in a limited number of subjects (MRI subgroup)
* Frequency of increase of liver enzymes according to World Health Organization (WHO) II criteria

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have given written informed consent prior to any trial related activities. Trial related activities are any procedures that would not have been performed during normal management of the subject
* Subjects with stable disease without relapses in the last 30 days
* Subjects aged between 18 and 55 years (both included)
* Subjects who suffer from definite RRMS according to Poser criteria (clinical definite multiple sclerosis [CDMS] or laboratory supported definite multiple sclerosis [LSDMS]) or definite MS according to McDonald criteria
* Subjects who have started treatment with Rebif® 44 mcg 3 months ago (+/- 1 month) including the titration phase
* Subjects who have a disability equivalent to an EDSS of 5.5 or less
* Subjects who have shown clinical activity defined as at least 1 documented relapse within the last year (A documented relapse is defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, persisting for more than 48 hours and with a previous period for more than 30 days with a stable or an improving condition. The exacerbation must be equivalent to an increase of at least 1 point in 2 functional systems or to an increase of 2 points in 1 system, either in the pyramidal, cerebellar, brain-stem, sensory, bowel and bladder, visual, cerebral or other functional system or an increase of at least half a point on the EDSS. Changes in bowel and bladder or cerebral functions should not solely be responsible for documentation of a relapse. The relapses must have been evaluated by a neurologist, retrospectively if necessary)
* Subjects must be prepared to and considered able to follow the protocol during the whole trial period and to attend the planned visits, even if the treatment has to be withdrawn
* Female subjects must either: be post-menopausal or surgically sterilized; or use a hormonal contraceptive or intra-uterine device (only following contraceptives are allowed: birth control pills, intra-uterine device, depot injection of gestagen, subdermal implant, hormonal vaginal ring and transdermal depot patches); or be sexually inactive for the duration of the study, and be neither pregnant nor breast-feeding (confirmation that the subject is not pregnant must be established by a negative serum human chorionic gonadotropin (hCG) pregnancy test within 28 days of Study Day 1 and a negative urine pregnancy test on Study Day 1. A pregnancy test is not required if the subject is post-menopausal or surgically sterilized)

Exclusion Criteria:

* Subjects with any condition that might give rise to similar symptoms as MS
* Subjects who have received any other immunomodulatory or immunosuppressive treatment 6 months prior to inclusion into the trial (the obligatory pre-study 3 months [+/- 1 month] period of Rebif® treatment not included)
* Subjects who have received mitoxantrone or total lymphoid radiation at any time
* Subjects who have received treatment with glucocorticoids or adrenocorticotropic hormone (ACTH) later than 1 month prior to inclusion into the trial
* Subjects who have experienced a relapse within 1 month prior to inclusion into the trial
* Subjects who have suffered from major depression
* Subjects with alcohol or drug dependency
* Subjects with cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmias, unstable or advanced ischemic heart disease (New York Heart Association [NYHA] grade III or IV), or significant hypertension (Blood Pressure > 180/110 millimeter of mercury [mmHg])
* Subjects with renal insufficiency defined as serum creatinine > 1.5 times the upper normal reference limit
* Subjects with alanine aminotransferase (ALAT) and asparagine aminotransferase (ASAT) (or either 1 if only 1 of the 2 is measured) levels more than 2 times the normal upper reference limit.
* Subjects with leucopoenia < 2500 per microliter (microL) or thrombopenia < 100000 per microL
* Subjects with any medical illness requiring treatment with systemic corticosteroids
* Subjects with any systemic disease that can influence the subject's safety and compliance, or the evaluation of the disability
* Female subjects who are pregnant or breastfeeding or who plan to become pregnant during the study
* Subjects with known or suspected allergy to minocycline or other tetracyclines
* Subjects who have participated in any other studies, involving other investigational products, within 30 days prior to participating in this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 305 (Actual)
Dates: Start 2006-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Soelberg Sørensen, Professor, Principal Investigator — Rigshospitalet,Blegdamsvej 9, 2100 København Ø, Scleroseklinikken afsnit 2082
Locations (1):
- Scleroseklinikken afsnit 2082, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One out of 305 participants was randomized by mistake and did not receive study medication.
Groups:
- Rebif®+ Minocycline: Participants who self-administered Rebif® (interferon beta-1 alpha [IFN beta-1a]) 44 microgram (mcg) as subcutaneous (sc) injection thrice weekly also received minocycline 100 milligram (mg) tablet twice daily as an add-on therapy in accordance with clinical practice for 96 weeks.
- Rebif® + Placebo: Participants who self-administered Rebif® (IFN beta-1a) 44 mcg as sc injection thrice weekly also received placebo tablets twice daily for 96 weeks.
Period: Overall Study
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Started | 149 (Number of participants treated.) | 155 (Number of participants treated.)
Completed | 80 | 88
Not Completed | 69 | 67
Not completed — Adverse Event | 47 | 31
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 3 | 5
Not completed — Lack of Efficacy | 2 | 12
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Planning to become pregnant/pregnancy | 1 | 0
Not completed — Other | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo | Total
Number analyzed (Participants) | 149 | 155 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.8) | 37.7 (8.6) | 37.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 102 | 198
  Male | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced First Documented Relapse
Description: Documented relapse: development of new/exacerbation of existing neurological symptoms, persisting for >48 hrs and with previous period for >30 days with stable/improving condition. Exacerbation = at least (>=)1 point increase in 2 functional systems/2 points increase in 1 system,either in pyramidal, cerebral, brain-stem, sensory, bowel and bladder, visual, cerebral or other functional system or >=0.5 point increase on expanded disability status scale (EDSS) which assesses disability in 8 functional systems with overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]).
Time Frame: Baseline up to 96 weeks (+/- 1 week) or early termination (ET)
Population: The Intention to Treat (ITT) population included all the participants who were randomized and received study medication.
Measure: Number; unit: participants
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 149 | 155
participants | 32 | 39

2. Secondary Outcome: Number of Participants With Documented Relapses
Description: Documented relapse: development of new/exacerbation of existing neurological symptoms, persisting for >48 hrs and with previous period for >30 days with stable/improving condition. Exacerbation was >=1 point increase in 2 functional systems /2 points increase in 1 system, either in pyramidal, cerebral, brain-stem, sensory, bowel and bladder, visual, cerebral or other functional system or >=0.5 point increase on EDSS which assesses disability in 8 functional systems with overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: ITT population included all the participants who were randomized and received study medication.
Measure: Number; unit: participants
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 149 | 155
participants
  0 | 117 | 116
  1 | 27 | 29
  2 | 2 | 9
  3 | 2 | 0
  4 | 1 | 1

3. Secondary Outcome: Number of New or Enlarging Lesions on Time Constant 2 (T2) Weighted Magnetic Resonance Imaging (MRI)
Description: Inflammatory disease activity was assessed by MRI measurement of the number of new or enlarging T2 lesions.
Time Frame: Final visit (96 weeks [+/- 1 week]) or ET
Population: Sub-group of ITT population included limited number of participants at pre-selected sites selected on basis of availability of MRI scanning facilities and the willingness of the site to participate.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 23 | 27
lesions | 3.0 (3.3) | 3.0 (4.6)

4. Secondary Outcome: Changes in Brain Volume Measured on Magnetic Resonance Imaging (MRI)
Description: Changes in brain volume were measured as the brain parenchymal fraction using MRI scans.
Time Frame: Screening , final visit (96 weeks [+/- 1 week]) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 23 | 26
cubic millimeter (mm^3) | -2997.4 (25799.3) | 5834.9 (20809.4)

5. Other Pre Specified Outcome: Number of Participants With Onset of Disability Progression
Description: Disability progression was defined as an increase, compared to baseline evaluation of >= 1.0 points on EDSS if EDSS was >= 1.0 at baseline or >=1.5 point on EDSS if EDSS was 0.0 at baseline. EDSS assesses disability in 8 functional systems with overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: ITT population included all the participants who were randomized and received study medication.
Measure: Number; unit: participants
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 149 | 155
participants | 6 | 3

6. Other Pre Specified Outcome: Number of Time Constant 2 (T2) Active Lesions
Description: Inflammatory disease activity was assessed by MRI measurement of the number of T2 active lesions.
Time Frame: Week 48 up to Week 96 (+/- 1 week) or ET
Population: Data was not analyzed due to insufficient number of participants available for the analysis of this measure and the study was prematurely terminated.
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Percentage of Time Constant 2 (T2) Active Scans Per Participant
Description: Inflammatory disease activity was assessed by MRI measurement of the percentage of T2 active scans.
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: as for outcome 6
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Burden of Disease
Description: The burden of disease (BOD) is the total area of MS lesions (abnormal plaques) in the brain measured on Time Constant 1 (T1) or T2 weighted MRI.
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: square millimeter (mm^2)
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 23 | 27
square millimeter (mm^2)
  Total area of lesions on T1 weighted MRI | 1599.4 (3196.3) | 1716.8 (2145.5)
  Total area of lesions on T2 weighted MRI | 4813.9 (8385.5) | 5717.3 (6587.0)

9. Other Pre Specified Outcome: Relapse Count
Description: A relapse was defined as the development of new or the exacerbation of existing neurological symptoms or signs, in the absence of fever, persisting for more than 48 hours and with a previous period for more than 30 days with a stable or an improving condition.
Time Frame: Week 48 (+/- 1 week) or ET
Population: Data was not analyzed due to insufficient number of participants available for the analysis of the measure and the study was prematurely terminated.
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Number of Relapse Free Participants Without Progression
Description: Analysis based on documented relapses (relapse: development of new/exacerbation of existing neurological symptoms, persisting for >48 hrs and with previous period for >30 days with stable/improving condition; relapse documented by exacerbation >=1 point increase in 2 functional systems/2 points increase in 1 functional system, or >=0.5 point increase on EDSS which assesses disability in 8 functional systems with overall score ranging from 0 [normal] to 10 [death due to MS]) and overall relapses (documented and undocumented relapses); undocumented relapses only fulfilled condition for relapse.
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: ITT population included all the participants who were randomized and received study medication. Number of participants analyzed "N" included those participants who were evaluated for this particular measure.
Measure: Number; unit: participants
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 141 | 147
participants
  Relapse free participants (documented relapse) | 105 | 108
  Relapse free participants (overall relapse) | 96 | 89

11. Other Pre Specified Outcome: Number of Participants With Total Number of Reported Relapses (Documented and Undocumented Relapses)
Description: Documented relapses (relapse: development of new/exacerbation of existing neurological symptoms, persisting for >48 hrs and with previous period for >30 days with stable/improving condition; relapse documented by exacerbation >=1 point increase in 2 functional systems/2 points increase in 1 functional system, or >=0.5 point increase on EDSS which assesses disability in 8 functional systems with overall score ranging from 0 [normal] to 10 [death due to MS]) and undocumented relapses only fulfilled condition for relapse.
Time Frame: Baseline up to 96 weeks (+/- 1 week) or ET
Population: ITT population included all the participants who were randomized and received study medication.
Measure: Number; unit: participants
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 149 | 155
participants
  0 | 107 | 96
  1 | 30 | 38
  2 | 6 | 17
  3 | 4 | 3
  4 | 1 | 0
  5 | 1 | 1

12. Other Pre Specified Outcome: Relapse Severity Based on Expanded Disability Status Scale (EDSS)
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. EDSS progression was defined as increase by at least 1 point if last value of EDSS was equal to 5.5 and by at least 0.5 points if last EDSS was more than 5.5.
Time Frame: 96 weeks (+/- 1 week) or ET
Population: ITT population included all the participants who were randomized to study medication. Number of participants analyzed "N" included those participants who were evaluated for this particular measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Number analyzed (Participants) | 125 | 136
Units on a scale | 1.90 (1.38) | 2.02 (1.42)

ADVERSE EVENTS:
Time Frame: Baseline to Week 100 (+/- 1 week) or ET.
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Rebif®+ Minocycline | Rebif® + Placebo
Serious Adverse Events (participants affected / at risk) | 11/149 | 21/155
Other Adverse Events (participants affected / at risk) | 51/149 | 35/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif®+ Minocycline (N=149) | Rebif® + Placebo (N=155)
Syncope (Nervous system disorders) | 1 | 1
Hypoesthesia (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abscess drainage (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Plastic surgery (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Transplant (Surgical and medical procedures) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depressive delusion (Psychiatric disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif®+ Minocycline (N=149) | Rebif® + Placebo (N=155)
Diarrhea (Gastrointestinal disorders) | 13 | 7
Nausea (Gastrointestinal disorders) | 22 | 7
Influenza like illness (General disorders) | 9 | 6
Nasopharyngitis (Infections and infestations) | 7 | 11
Hepatic enzyme increased (Investigations) | 6 | 8
Dizziness (Nervous system disorders) | 9 | 2
Headache (Nervous system disorders) | 13 | 15
Depression (Psychiatric disorders) | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other